CLINICAL TRIAL: NCT03945162
Title: A Phase II Clinical Study of Intravesical Ruvidar® in Patients With BCG-Unresponsive Non-Muscle Invasive Bladder Cancer ("NMIBC") Carcinoma In-Situ ("CIS") or Patients Who Are Intolerant to BCG Therapy ("Study II")
Brief Title: Intravesical Photodynamic Therapy ("PDT") in BCG-Unresponsive/Intolerant Non-Muscle Invasive Bladder Cancer ("NMIBC") Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Theralase® Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruvidar® (TLD-1433) NMIBC PDT
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Non-Muscle Invasive Bladder Cancer ("NMIBC") Unresponsive/Intolerant to BCG
Keywords: Photodynamic Therapy; Non-muscle invasive bladder cancer ("NMIBC"); Urothelial carcinoma; Ta bladder cancer; T1 bladder cancer; Unresponsive/Intolerant to BCG
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- 0.70 mg/cm^2 Ruvidar® (TLD-1433) Bladder instillation and Photodynamic Therapy (Experimental): Each Study Procedure is a single instillation of Ruvidar® (TLD-1433) (at the therapeutic dose of 0.70 mg/cm^2) will be infused intravesically into the bladder for approximately 60 minutes, followed by PDT treatment using the TLC-3200 system, which is performed after Ruvidar® (TLD-1433) has been rinsed from the bladder. One Study Procedure will be performed, with up to 2 additional re-induction Study Procedures based on patient response.
  Interventions: Combination Product: Ruvidar® (TLD-1433) bladder infusion and PDT

INTERVENTIONS:
Combination Product: Ruvidar® (TLD-1433) bladder infusion and PDT — Ruvidar® (TLD-1433) is infused into the bladder and treatment of bladder wall with PDT light activation using the TLC-3200 system.

SUMMARY:
This is a phase II, open-label, single-arm, multi-center Study conducted in Canada and the United States. Patients with Non-Muscle Invasive Bladder Cancer ("NMIBC") Carcinoma In-Situ ("CIS") (with or without resected papillary disease (Ta, T1)) that are considered Bacillus Calmette-Guerin ("BCG")-Unresponsive or who are intolerant to BCG therapy. BCG-Unresponsive is at least one of the following: At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy; or, at least five of six doses of an initial induction course plus at least two of six doses of a second induction course. Patients experiencing disease relapse within 12 months after finishing the second course of BCG therapy are considered BCG-Unresponsive. The Study will consist of 90 patients who will undergo one (1) Study Procedure, with up to two (2) additional re-induction Study Procedures based on patient response.

DETAILED DESCRIPTION:
1. Overall Study Design and Plan: Description

   This is a phase II, open-label, single-arm, multi-center Study conducted in Canada and the United States. Patients with NMIBC CIS (with or without resected papillary disease (Ta, T1)) that are considered BCG-Unresponsive or are intolerant to BCG therapy that meet the inclusion and exclusion criteria will be enrolled and treated. The Study will consist of 90 patients who will receive one (1) Study Procedure, with up to two (2) additional re-induction Study Procedures based on patient response.
2. Screening Period

   Patients will be qualified for Study II entry by review of inclusion and exclusion criteria during the Screening Period, which will last up to 60 days.
3. Follow-Up Phase

   All patients enrolled and treated by the treatment procedure will be followed until the End of Study defined as completion of all required assessments after 15 months of follow-up post primary study treatment or due to early discontinuation or withdrawal of informed consent.

   During the Follow-Up Phase, information on efficacy and safety will be collected. Assessments will be conducted at Day 0, 7, 90, 180, 270, 360 and 450 days.

   Survival surveillance for all patients who achieve a CR or Indeterminate Response ("IR") (negative cystoscopy and positive urine cytology, without confirmatory negative bladder cancer biopsies) at four hundred and fifty (450) days and remain in Study II will be monitored for up to one thousand and eighty (1080) days post primary Study II Treatment, recording: efficacy, safety and incidence of radical cystectomy every ninety (90) days for the first seven hundred and twenty (720) days, then every one hundred and eighty (180) days, until one thousand and eighty (1080) days.
4. Study Drug and PDT Administration

Ruvidar® (TLD-1433) for intravesical administration is supplied as a lyophilisate for suspension in Sterile Water For Injection ("SWFI") into the bladder and is packaged in the dark in amber USP Type III glass vials, which are stored at 3 to 8 degree Celsius. Up to 24 hours before administration, it is reconstituted with SWFI to obtain the final clinical dilution.

Ruvidar® (TLD-1433) will be supplied to each Study II site by Theralase®. Instillations cannot be done immediately following biopsy taken by Trans-Urethral Resection of Bladder Tumour ("TURBT"). Investigators must wait a minimum of 7 days before dosing patients after a TURBT/biopsy, and/or until any bladder wall integrity issues have resolved. Dose/volume reductions are not allowed during Study II.

Upon determination of the bladder volume (during the screening period) through a self-recorded voiding diary, Ruvidar® (TLD-1433) will be diluted with SWFI to the proper concentration. On day 0 (Primary Study Procedure day), patients will be asked to restrict fluid intake 12 hours before Study Drug instillation. Study Drug must be instilled into the patient's empty bladder. Before instillation, a regular transurethral catheter should be inserted and the bladder drained. A single instillation of Ruvidar® (TLD-1433) will be infused intravesically for approximately 60 minutes, followed by 1 wash with SWFI. The bladder will be distended using a second instillation of SWFI to prevent folds that may prevent uniform light illumination. The Computer Operator worksheet must be completed during the Study Procedure and data must be promptly transferred to the corresponding electronic Case Report Form ("eCRF") page.

The optical fiber with spherical diffuser will be positioned through the cystoscope in the geometric center of the bladder with the aid of TLC-3200 and will be locked into place using an endoscope holder for continuous irradiation for the total exposure time. The optical power and treatment time will be determined to provide the correct dose of laser light to the bladder surface area. Green laser light (wavelength = 532 nm, energy = 90 J/cm2) will be irradiated from the emitter optical fiber via the spherical diffuser.

4.1 Dosing Schedule

One Study Procedure is planned, with up to two additional re-induction Study Procedures based on patient response. Each Study Procedure is a single whole bladder intravesical Ruvidar® (TLD-1433) instillation followed by PDT with the TLC-3200 System.

4.2 PDT Disruption

Patients with persistent or recurrent NMIBC CIS alone (or with recurrent Ta/T1 (noninvasive papillary disease/tumour invades the subepithelial connective tissue)) disease within 12 months of completion of BCG therapy (BCG-Unresponsive) or who are intolerant to BCG therapy will be treated with this Protocol. If one or more papillary tumours are seen at the time of Study Treatment (maximum 12 weeks after TURBT), the patient will be resected via TURBT and will be treated with this Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide a written Informed Consent Form ("ICF") for the Study.
2. Be > 18 years of age on day of signing ICF.
3. Have histologically confirmed NMIBC CIS via biopsy with/without resected papillary disease (Ta, T1) (high grade) using the 2004 World Health Organization ("WHO") / International Society of Urologic Pathology classification system. The most recent cystoscopy / TURBT must have been performed within 12 weeks of the Study Procedure date to confirm: histology, grade and stage.
4. Intolerant to BCG or considered BCG-Unresponsive, which is at least one of the following:

   * At least five of six doses of an initial induction course, plus at least two of three doses of maintenance therapy, or
   * At least five of six doses of an initial induction course, plus at least two of six doses of a second induction course.
5. Are not candidates for cystectomy on medical grounds or refuse radical cystectomy.
6. Have an Eastern Cooperative Oncology Group ("ECOG") performance score of 0 to 2.
7. Have satisfactory bladder function. Ability to retain Study Drug for a minimum of 60 minutes.
8. Are available for the duration of the Study including follow-up (approximately 15 months).
9. Female patients of childbearing potential must have a negative Human Chorionic Gonadotropin ("HCG") pregnancy test taken during the screening visit and confirmed prior to the Study Procedure.
10. Female patients of childbearing potential must be willing to use 2 methods of birth control (i.e.: oral contraceptive, pills, diaphragm or condoms) or be surgically sterile, or abstain from heterosexual activity for two weeks after the Study Procedure. Patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.

Exclusion Criteria:

1. Past or current muscle invasive (i.e.: T2, T3, T4) or metastatic urothelial carcinoma.
2. Has concurrent extravesical (i.e.: urethra, ureter, renal pelvis, prostate or prostatic ducts) non-muscle invasive transitional cell carcinoma of the urothelium. (confirmed by staging to exclude extravesical disease, which may include radiological imaging and/or biopsy) within 3 months of enrollment:

   If previous work up occurred more than 3 months prior to enrollment, staging for extravesical disease must be repeated prior to enrolment in order to determine eligibility.
3. Active gross hematuria.
4. Have a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer or localized prostate cancer under active surveillance with Gleason 6 disease. A history of prostate cancer that was treated with definitive intent (surgically or through radiation therapy) is acceptable, provided that the following criteria are met: Stage T2N0M0 or lower Prostate-Specific Antigen ("PSA") undetectable for 2 years while off androgen deprivation therapy or no more than 2 consecutive rising PSAs.
5. Have a history or current evidence of any condition, therapy, surgery or laboratory abnormality that, in the opinion of the PI, might confound the results of the study, interfere with the patient's participation in the study, or is not in the best interest of the patient to participate.
6. Currently receiving treatment with a prohibited concomitant therapy (refer to 12.2.1, Prohibited Medications).
7. Participated in a study with an investigational agent or device within 1 month from the first dose of current Study Procedure.
8. Prior treatment with an intravesical chemotherapeutic agent within 1 month of the first dose of current Study Drug, with the exception of a single perioperative dose of chemotherapy immediately post-TURBT (not considered treatment).
9. Have an active infection requiring systemic therapy, including active or intractable Urinary Tract Infection ("UTI"), not resolved prior to the procedure.
10. Has any contraindication to general or spinal anesthesia.
11. Is pregnant or breastfeeding within the projected duration of Study II, starting with the screening visit through to two weeks following the last Study Procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-08-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy, evaluated by Complete Response ("CR"). | Throughout Study II and up to the completion of the follow-up phase (15 month)
  The primary endpoint of Study II is efficacy, evaluated by the Complete Response ("CR") at any time point in patients with Carcinoma In-Situ ("CIS") with resected papillary disease.
  Patient CR is defined as at least one of the following:
  * Negative cystoscopy and negative (including atypical) urine cytology
  * Positive cystoscopy with biopsy-proven benign or low-grade NMIBC and negative cytology
  * Negative cystoscopy with malignant urine cytology, if urothelial cancer is suspected in the upper tract or prostatic urethra and random bladder biopsies are negative.

SECONDARY OUTCOMES:
Efficacy, evaluated by the duration of CR | Throughout Study II and up to the completion of the follow-up phase (15 month)
  Assessment of the Duration the CR is maintained after an initial CR is achieved.
Three year patient assessments, for observation only. | Follow-up phase from 15 to 36 months for those who remain in Study.
  Survival surveillance for all patients who achieve a CR or Indeterminate Response ("IR") (negative cystoscopy and positive urine cytology, without confirmatory negative bladder cancer biopsies) at four hundred and fifty (450) days and remain in Study II will be monitored for up to one thousand and eighty (1080) days post primary Study Procedure, recording: efficacy, safety and incidence of radical cystectomy every ninety (90) days for the first seven hundred and twenty (720) days, then every one hundred and eighty (180) days, until one thousand and eighty (1080) days.

OTHER OUTCOMES:
Safety, evaluated by the incidence and severity of Adverse Events. | Throughout the study and up to the completion of the follow-up phase (15 month)
  The tertiary endpoint of Study II is safety, evaluated by the incidence and severity of Adverse Events ("AEs"), Grade 4 or higher that do not resolve within 450 days post initial treatment; whereby: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening or disabling, Grade 5 = Death

CONTACTS AND LOCATIONS:
Overall Officials: Girish Kulkarni, MD, FRCSC, Principal Investigator — University Health Network, Toronto
Locations (16):
- United States (10):
  - Site 02-012 - University of Chicago, Chicago, Illinois
  - Site 02-016 - Urology of Indiana, Greenwood, Indiana
  - Site 02-015 - Associated Medical Professionals of New York, Syracuse, New York
  - Site 02-017 - Central Ohio Urology Group, Gahanna, Ohio
  - Site 02-008 - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Site 02-006 - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Site 02-007 - Urology Associates, P. C, Nashville, Tennessee
  - Site 02-010 - Urology San Antonio P. A, San Antonio, Texas
  - Site 02-009 - Virginia Urology, Richmond, Virginia
  - Site 02-011 - University of Wisconsin Health University Hospital, Madison, Wisconsin
- Canada (6):
  - Site 01-005 - The Vancouver Prostate Centre - Diamond Health Care Centre - Vancouver General Hospital, Vancouver, British Columbia
  - Site 01-004 - Nova Scotia Health Authority - Centre for Applied Urology Research, Halifax, Nova Scotia
  - Site 01-014 - St. Joseph's Healthcare, Hamilton, Ontario
  - Site 01-002- London Health Sciences Centre - Victoria Hospital, London, Ontario
  - Site 01-001 - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - Site 01-003 - McGill University Health Centre - Glen-Cedars Cancer Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No